CLINICAL TRIAL: NCT06508905
Title: The Effect of Sleep Companion Application on Psychosocial Symptoms in Hospitalized Children
Brief Title: Sleep Buddy Application in Hospitalized Children
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Medipol University Hospital (Other)
Responsible Party: Principal Investigator, aysel kokcudogan, Assistant Professor, Istanbul Medipol University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: E-76728045-806.01.03-226794342
Record Dates: First submitted 2024-07-15; First posted 2024-07-18 (Actual); Last update posted 2024-10-03 (Actual); Status verified 2024-10

CONDITIONS: Main Heading (Descriptor) Terms
Keywords: hospital; child; sleep companion; psychosocial symptoms

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sleep buddy (Experimental): Children who did not have their own sleeping companion were given a toy selected as a sleeping companion. The toy was introduced to the children and accompanied them for 3 days during their hospitalization.
  Interventions: Other: Sleep buddy
- control group (No Intervention): After the child in the control group was hospitalized in the clinic, routine hospitalization procedures were performed and no intervention was performed. The child was observed during the three days of hospitalization. It was observed that the children did not have their own toys with them.

INTERVENTIONS:
Other: Sleep buddy — The toy chosen as a sleep companion was introduced to the children in the experimental group and they were told that it would accompany them for 3 days during their hospitalization. Before giving the sleep companion, parents and children were informed about the sleep companion and their questions about the study were answered. Children who did not have their own sleep companion were included in the sample. The child was encouraged to sleep and spend time with the given sleep buddy and the family was also informed.
  Arms: Sleep buddy

SUMMARY:
The study was planned as a randomized controlled experimental study to investigate the effect of sleep companion application on psychosocial symptoms in hospitalized school children aged 6-12 years.

DETAILED DESCRIPTION:
The sample of the study consisted of a total of 97 school-age children hospitalized in the Pediatrics and Pediatric Surgery-Endocrine Service of the Health Services Application and Research Hospital of a university hospital and in the Pediatrics Service of a state hospital. Children who met the inclusion criteria and whose written and verbal consent was obtained from their parents for participation in the study after being informed were included in the study.

The study was completed as 50 control and 47 experimental group with 3 missing persons in the experimental group.

Data were collected using the "Introductory Information Form" and "Psychosocial Symptoms Diagnostic Scale for Hospitalized Children (PSDS)" tools.

The toy, which was selected as a sleep companion for the children in the experimental group, was introduced to the children and accompanied them for 3 days during their hospitalization. The experimental and control groups were observed for psychosocial symptoms.

The data will be analyzed with SPSS software.

ELIGIBILITY:
Inclusion Criteria:

* Hospitalized school-age children (6-12 years old),
* No mental disability,
* Volunteer to participate in the research,
* No allergies,
* Children who are hospitalized for at least 3 days

Exclusion Criteria:

* Hospitalized children under 6 years of age and over 12 years of age,
* Predicted discharge in less than 3 days,
* Children with a sleeping companion

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 97 (Actual)
Dates: Start 2023-06-01 (Actual); Primary Completion 2024-01-30 (Actual); Study Completion 2024-10-30 (Estimated)

PRIMARY OUTCOMES:
Psychosocial symptoms diagnostic scale | Used 3 days after the sleep companion app. The scale administration took 15 minutes.
  Determination of psychosocial symptoms of hospitalized children The highest score that can be obtained from the scale is "48" and the lowest score is "0". A high score on the scale means that the hospitalized school child has psychosocial problems.

CONTACTS AND LOCATIONS:
Overall Officials: Aysel Kokcu Dogan, Ph.D, Study Director — Medipol University
Locations (1):
- Medipol University, Istanbul, Beykoz, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No